CLINICAL TRIAL: NCT03385278
Title: Effects of Repetitive Transcranial Magnetic Stimulation on the Disorders of Consciousness
Brief Title: Transcranial Magnetic Stimulation in Patients With Disorders of Consciousness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TMS
Record Dates: First submitted 2017-10-24; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-10

CONDITIONS: Disorder of Consciousness
Keywords: TMS;DOC
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: This study was designed and performed as a randomized, controlled cross-over trial. All patients were randomly received active 20-Hz rTMS and sham stimulation for 5 consecutive days, in separate sessions spaced one week.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-sham (Experimental): the group first received real rTMS,then sham one.
  Interventions: Other: rTMS
- sham-real (Experimental): the group first received sham rTMS,then real one.
  Interventions: Other: rTMS

INTERVENTIONS:
Other: rTMS — 20HZ Repetitive Transcranial Magnetic Stimulation

SUMMARY:
Transcranial magnetic stimulation involves the use of alternating magnetic fields to stimulate neurons in the brain.To date, several studies have focused on the use of TMS in patients with impaired consciousness.However,its therapeutic effects have been variously documented.So,in this study ,investigators explore the effects of rTMS with cross-over design.

DETAILED DESCRIPTION:
Background:Repetitive transcranial magnetic stimulation (rTMS) was supposed as an experimental approach to disorders of consciousness treatment. Its therapeutic effects have been variously documented.

Objective: The study aimed to investigate the reactivity of electroencephalography (EEG) and the clinical response of patients with disorders of consciousness and explore the neuromodulatory effects of high-frequency rTMS in DOC.

Method:In this randomised,sham-controlled study,real or sham 20 Hz rTMS were applied to the left primary motor cortex (M1) of participants with disorders of consciousness for 5 consecutive days . Evaluations were blindly performed at baseline, immediately after the end of the 5-days treatment and 1 week later with the JFK Coma Recovery Scale-Revised (CRS-R) scale and EEG.

Hypothesis:Real rTMS can be an effective awakening method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 14 to 65 years old;
2. no centrally acting drugs;
3. no neuromuscular function blockers and no sedation within the prior 24 hours; 4.periods of eye opening (indicating preserved sleep-wake cycles);

5.DOC patients, including vegetative state and minimally consciousness state.

Exclusion Criteria:

1. History with nervous or spirit disorders, or some other serious diseases such as cardiac or pulmonary problems;
2. with a contraindication for rTMS

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-04 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
the JFK Coma Recovery Scale-Revised (CRS-R) scale | at baseline (T0), immediately after the end of the 5-day treatment (T1), 1 week later (T2).Investigators observed the changes from baseline to the end of stimulation.
  The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors.

SECONDARY OUTCOMES:
EEG data ( electrophysiological parameters) | at baseline (T0), immediately after the end of the 5-day treatment (T1), 1 week later (T2)
  delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz) and beta (12-30 Hz).an increase of delta and theta activity usually reflects encephalopathy and/or structural lesions, interpreted as poor outcome predictor of DOC .The power of α and β is related to the chance of recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- Hangzhou Hospital of Zhejiang CAPR, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cincotta M, Giovannelli F, Chiaramonti R, Bianco G, Godone M, Battista D, Cardinali C, Borgheresi A, Sighinolfi A, D'Avanzo AM, Breschi M, Dine Y, Lino M, Zaccara G, Viggiano MP, Rossi S. No effects of 20 Hz-rTMS of the primary motor cortex in vegetative state: A randomised, sham-controlled study. Cortex. 2015 Oct;71:368-76. doi: 10.1016/j.cortex.2015.07.027. Epub 2015 Aug 4. PMID 26301875
- [Derived] He F, Wu M, Meng F, Hu Y, Gao J, Chen Z, Bao W, Liu K, Luo B, Pan G. Effects of 20 Hz Repetitive Transcranial Magnetic Stimulation on Disorders of Consciousness: A Resting-State Electroencephalography Study. Neural Plast. 2018 Mar 25;2018:5036184. doi: 10.1155/2018/5036184. eCollection 2018. PMID 29770146